CLINICAL TRIAL: NCT04196556
Title: Effectiveness of an Intervention Programme (FAMILIAS ACTIVAS) for Childhood Obesity: Cluster Randomized Controlled Trial
Brief Title: Effectiveness of an Intervention Programme for Childhood Obesity: FAMILIACT
Acronym: FAMILIACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Diego José Villalvilla Soria, Nurse. Clinical research, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI 25/17
Record Dates: First submitted 2019-12-02; First posted 2019-12-12 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Primary Health Care; Nursing intervention; Family educational intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: A multicenter Cluster Randomized Clinical Trial
Masking Description: Intervention can't be masked. Statistician conducting the analysis will not know to which study arm a given patient has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Families (Experimental): Usual care plus intervention active families. This intervention, based on the methodology of meaningful learning, will have two components: group education directed to parents (caregivers) and education directed to children in the reviews in consultation. The group intervention will consist of 6 sessions, with a biweekly / monthly frequency, will be taught as determined in the program monitoring annex, in the 3 months after the initial assessment. The content of the sessions is defined in attached annex. Regarding the proposed methodology, it has nuances and tools different from the traditional ones to achieve significant learning in the field of health. It is based on participatory methods and a more profound modification of knowledge, skills, emotions and attitudes than the brief advice that is used in family intervention in scheduled consultations.
  Interventions: Behavioral: Active Families; Other: Madrid's Primary Healthcare Standardized Service portfolio
- Control group (Active Comparator): Usual care:
  The activities included in the Service for Attention to Patients with Childhood Obesity will be carried out in the Madrid's Primary Healthcare Standardized Service portfolio, which establishes a monthly follow-up in the first 6 months and bimonthly of month 6 to 12. To this At least the child and the primary caregiver, the child's educational agent, will be consulted and will receive support documentation to exercise and reinforce their role.
  Interventions: Other: Madrid's Primary Healthcare Standardized Service portfolio

INTERVENTIONS:
Behavioral: Active Families — This intervention, based on the methodology of meaningful learning, will have two components: group education aimed at parents (caregivers) and and education directed to children in the reviews in consultation. Group education (caregivers) groups will consist of 6 sessions, which will be given every two weeks, as determined in the program's follow-up annex, in the 3 months after the initial assessment. The content of the sessions is defined in attached annex. Regarding the proposed methodology, it has nuances and tools different from the traditional ones to achieve significant learning in the field of health. It is based on participatory methods and a more profound modification of knowledge, skills, emotions and attitudes than the brief advice that is used in family intervention in scheduled consultations.
  Other Names: Madrid's Primary Healthcare Standardized Service portfolio
  Arms: Active Families
Other: Madrid's Primary Healthcare Standardized Service portfolio — An anamnesis or functional assessment on the following aspects:
  o Family history of obesity up to 2nd degree inbreeding. o Nutritional status - metabolic that includes at least no meals/day and daily consumption of liquids, fruits, vegetables, dairy, fats and sugars. o Activity - exercise that includes at least the type and intensity of exercise and time spent on sedentary activities (television, video games or the like). o Self-concept that includes at least the existence or not of behavioral problems and body image problems. o Role - relationships that include at least the performance of extracurricular activities.
  A care plan in relation to identified problems and/or situations reviewed on a biannual basis.
  They will be supplemented with the study-specific variables listed in the data collection notebook.

SUMMARY:
Objectives. To assess the effectiveness of a programmed family/group intervention to reduce weight in the treatment of obesity in children 7 to 12 years old in front of usual treatment. Design. Cluster randomized controlled trial, multicenter. Location. Primary health care centers. Participants. Obese children 7 to 12 years old of primary health care centers. Body mass index (BMI) > P 97. Patients give Informed consent. Sampling. Randomized cluster assigned. Assignation unit: primary care center. Analysis unit. Patient (Children and childminder). Size: 280 patients (140 by group). Principal measurements Variables.BMI z score (BMI-SDS) after the 6 month intervention and after 12 -month follow-up. Secondary Measurements Variables. quality of Mediterranean diet, Brief questionnaire of physical activity in children. Brief Physical Activity Assessment Tool (BPAAT) for adults (Parents) , apgar-family questionnaire. sociocultural level., educational level, Gender. Age. BMI parents, family antecedent. Analysis: Primary effectiveness. Initial comparability of groups according to the outcome and confusion variables. Mean differences in z score of BMI with 95% confidence intervals, between groups and generation of a multivariate and multilevel model. Analysis by intention to treat.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effectiveness of a family intervention to reduce obesity in children. Overweight and obesity, as defined by the World Organization of Health (WHO) as abnormal or excessive fat accumulation that can be harmful to health, they are considered by this body as one of the most important public health problems of the century XXI, which is the fifth leading death risk factor in the world.

OI has been associated with high co-morbidity in adulthood. The percentile increase in body mass index (BMI) in OI increases the incidence of cases of hypertension , dyslipidemia, left ventricular hypertrophy, atherosclerosis, metabolic syndrome, type 2 diabetes, sleep disorders, as well as psychological effects, such as stigmatization, discrimination, depression and emotional trauma. Obesity in childhood also substantially increases the risk of being an obese adult. In addition, childhood obesity is an independent risk factor for obesity in adulthood. Criteria favorable to therapeutic intervention in cases of obesity are based on the demonstration that with a moderate weight loss (5-10%) can achieve a marked improvement in the associated comorbidity and quality of life even in severe obesity. The prevalence of multiple risk factors increases as the BMI percentile increases, and severe obesity is associated with an increased risk of comorbidity and resistance to sustained weight loss.

The discussion about the relevance and form of the approach to childhood obesity is an open and current issue. A 2007 Cochrane review established that there may be a benefit to behavioral treatment where parents are given responsibility for behavioral change and this is done as a family. To start the intervention, professionals with specific training in physical activity and nutrition applied in childhood, behavioral intervention techniques and promotion of healthy habits in working with families are required.

Another more recent review focused on evaluating the effectiveness of different interventions to treat childhood obesity concludes that although there is not much quality data to recommend a treatment program superior to another, the combined lifestyle and behavior interventions in Comparison with standard care or self-help can lead to a significant reduction in overweight in children and adolescents.

Another aspect to take into account is the relevance of the early intervention of obesity during childhood-adolescence, since it is at this stage that the eating habits and practice of physical exercise are consolidated, in addition to where they conform the personality characteristics of the individual.

The family intervention is proposed as one of the areas most likely to be successful in treating childhood obesity. There are several clinical trials that evaluate different interventions aimed primarily at families and show that they have beneficial effects in the promotion of healthy behaviors related to food and exercise in boys and girls, in addition to highlighting the importance of a combined dietary, behavioral and physical activity component.

The few studies carried out in the specific field of community nursing have small sample sizes and have not shown that the intervention in nursing consultation has been effective as far as weight loss is concerned. Another study comparing the effect of medical counseling and group therapy in childhood obesity concluded that cognitive behavioral therapy is more effective than medical advice and that none of the two treatment improved results compared to the untreated group. There are several limitations that could justify this result, among others the possible insufficient family involvement that is considered of vital importance.

4. 1. CONCEPTUAL Hypothesis : The "Active Families" intervention program is more effective than the usual practice to reduce the weight of children from 7 to 12 years old with obesity at the end of the intervention and at 6 and 12 months after the start of the intervention.

4.2. OPERATIONAL HYPOTHESIS: The "Active Families" family intervention program decreases an average of 0.5 standard deviations plus the BMI of children with childhood obesity than the usual practice at the end of the intervention and at 6 and 12 months after the start of the intervention.

4. 3.OBJECTIVES Main objective: To evaluate the effectiveness of a family intervention program to reduce weight in children aged 7 to 12 years with childhood obesity compared to the usual practice at 6 and 12 months after the intervention.

Secondary Objectives:

1. Evaluate the effectiveness of a family intervention program aimed at children aged 7 to 12 with childhood obesity to improve the quality of food.
2. Evaluate the effectiveness of a family intervention program aimed at children aged 7 to 12 with childhood obesity to increase physical activity.
3. Evaluate the effectiveness of a family intervention program aimed at children aged 7 to 12 with childhood obesity to increase the physical activity of the main caregiver.

Design : Controlled clinical trial with randomized allocation by conglomerates, open, multicenter, 12 months follow-up, in primary care consultations. Location or scope: Health Centers of the Community of Madrid. Duration: 12 months years. Study population : Children diagnosed with obesity attended in primary care consultations of 7 to 12 years of both sexes.

Sample size: It has been estimated for a difference of 0.5 standard deviations ( clinically relevant result ), and a power of 80%. Specifying a total of 170 children, 85 in each group. Correcting for a design effect of 1,369, considering an ICC of 0,041 (28) and an average cluster size of 10 boys or girls, 233 boys or girls are required. Estimating losses of 20%, the final size is 280 children, 140 in each group. Sampling : Randomized allocation by conglomerates (nurses). Randomization unit: Primary Health Care Centers. The Health Centers will be assigned to the intervention or to the control group through a random sequence generated by computer. Analysis Unit: Diads child / caregiver. They will be included by consecutive sampling. During the consultation, that child susceptible to being included in the study will be informed and offered participation. If you agree to participate, you will be asked to complete and sign the informed consent and verify that you meet all the inclusion criteria and none of the exclusion criteria. Randomization of health centers will be carried out once the eligible dyads have been selected for the study, so that the recruitment by professionals is not influenced by the branch of the study to which they have been assigned.

Data Collection :

The information will be collected through clinical interview and physical examination and the data will be recorded in an electronic data collection notebook specially designed for this study. The variables will be collected during 4 visits: at the beginning of the study, at the end of the intervention, at 6 and 12 months.

Losses in participation: Losses and abandonment of follow-up during the study. The cause will be collected (voluntary abandonment, displacement, comorbidity, death and cause). If a patient does not attend a session, at least two telephone contact attempts will be made.

Control group . The activities included in the Service for Childhood Obesity Patients of the Portfolio of Standardized Primary Care Services of the Community of Madrid will be carried out , which establishes a monthly follow-up in the first 6 months and bimonthly from 6 to 12. This consultation will be attended by at least the child and the primary caregiver, the child's educating agent, and will receive supporting documentation for Exercise and strengthen your role.

* Experimental group : Regular intervention plus intervention active families. This intervention, based on the methodology of meaningful learning , it will have two components: group education aimed at parents (caregivers) and education aimed at children in the reviews in consultation. The group intervention will consist of 6 sessions, which with a biweekly / monthly frequency, will be taught as determined in the program monitoring annex, in the 3 months after the initial assessment.

In order to normalize and protocolize the activities in both groups (intervention and control) a training session will be held prior to the start of the field work

Analysis Strategy :

It will be done according to the intention to treat principle.

1. Review of the data and descriptive analysis of the study variables evaluating the normality of the distribution with its corresponding 95% confidence intervals .
2. Initial comparability of the groups according to the outcome and confusion variables . Chi square test for qualitative variables and used the T of Student for quantitative (if they conform to a normal distribution) or nonparametric test (if not follow a normal distribution).
3. Principal effectiveness analysis: calculation of the difference in means of the Z Score between groups, together with their 95% Confidence Interval.
4. To assess the effect of the intervention on the Z score of the BMI, a multivariate analysis will be carried out using a mixed multilevel model (level 1: child / caregiver dyad ; level 2: professional dyad / health center), with the intervention as fixed effects factor and professionals or centers as random effects factor (Brown H and Prescott R (1999). Applied mixed models in medicine. New York: Wiley.).

This same analysis will be applied to analyze the impact of the intervention on the rest of the quantitative dependent variables contemplated in the secondary objectives of the study.

1. - Technical Group.

   * Preparation of the Guide to Attention to Sedentary and Childhood Obesity (Educational Materials of Active Families).
   * Childhood Obesity Care Program (Standardization of the usual service portfolio process in which the standardized care plan for childhood obesity is also included). Presentation of the same to the professionals assigned to the control group through a clinical session of two hours of training.
   * Design of electronic Data Collection Notebook (CRD) accessible from the AP computer HC and a database containing CRD information
   * Periodic monitoring of the information collected: Evolution of patient acquisition and detection of recorded data errors, due to violation of the researcher's manual. For this, the contracted computer technicians will design specific SQL statements (Programming language).
   * Data debugging: validation process by searching for repeated records, and inconsistent, illogical or out of range values.
   * Bibliographic update and management of bibliographic references.
2. - Assistance Group: This group will be formed by nurses and pediatricians of the participating centers. There will be two people responsible for implementing the program in each center that will facilitate contact with the coordinating group. Perform the tasks of the assistance group:

   * Recruitment of patients and assess the inclusion criteria. Carry out the intervention assigned to the patients. Collection and registration of data in the CRD.
   * The professionals of the care group will appear as an attached note in the possible publications derived from the study, so that the names of all the participants appear in the bibliographic databases. Inclusion in these groups will depend on the involvement and activities carried out by each collaborator.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 7 and 12 years old.
* Obesity: defined by a BMI equal to or greater than P97 for age and sex in the curves and growth charts of the semilongitudinal study by Hernández (1988). Definition recommended by the Clinical Practice Guide of the Ministry of Health. To have primary caregiver.
* Be able to follow the demands of the trial (child and primary caregiver participants).
* Have no intention of moving in the following 12 months. Give informed consent to participate in the study.

Exclusion Criteria:

* Intention of moving in the following 12 months.
* Do not sign informed consent.
* Sensory, psychiatric or occupational limitations of caregivers that do not allow follow-up sessions.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 253 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Change Score Z score of the BMI of the child | 4, 6 and 12 months from the start of the intervention using the tables of Hernández 1988
  Change Score Z score of the BMI at the end of the intervention and at 4, 6 and 12 months from the start of the intervention using the tables of Hernández 1988 (annex 8). The Z score of the BMI is the variable of choice according to international proposals to explain the changes related to sex and age over time after an intervention in childhood obesity (12). Calculation of the score Z score of the BMI = (X-X') / DS. In which X = BMI of the child, X '= average BMI value for a specific age and sex according to the 1988 Hernández tables and SD = standard deviation of the mean BMI value according to the 1988 Hernández tables.
Weight of the child | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment.
  Weight in kilograms
Height of the child | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment.
  height in meters
BMI of the child | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment.
  weight and height will be combined to report BMI in kg/m^2)

SECONDARY OUTCOMES:
KIDMED test. Quality of the diet | Baseline (at the start of the intervention) and at 12 months of treatment
  KIDMED test consisting of 16 issues that are based on the principles of the Mediterranean Diet. The score that can be achieved after answering the questions of the test goes from O to 12 and allows to make a classification of the quality of the diet in three groups: <_3 poor quality, 4-7 average quality and >8 optimal quality.
Physical activity of the child (Gasol Foundation Questionnaire for assessment of physical activity and sedentary lifestyle adapted version ) | Baseline (at the start of the intervention) and at 12 months of treatment
  Physical activity questionnaire adapted version . It measures physical activity, PAU QUESTIONARY, allows to classify as active/inactive ; sedentary/non-sedentary physical exercise and sedentary leisure. The questions of which allow researchers to know whether or not children meet the recommendation of the World Health Organization (WHO) to do a minimum of 60 minutes of physical activity per day. Complying with the recommendation determines that the child is ACTIVE. Failure to comply with the recommendation classifies the child as inactive. Two questions value if you accumulate 2 hours a day on a regular basis of sedentary leisure (screens). Regularly accumulating more than 2 hours classifies the child as sedentary, not reaching the two hours of daily sedentary leisure classifies the child as nonsedentary.
  The questionnaire classifies boys and girls according to the minutes of exercise accumulated per week
Family Function. APGAR FAMILIAR | Baseline (at the start of the intervention) and at 12 months of treatment.
  Application to the main caregiver of the Apgar-family questionnaire that has demonstrated its validity and reliability in primary care. APGAR FAMILAR.
  There are five questions, each question is scored on a value from 0 to 2, eventually getting an index of 0 and 10.
  Interpretation:
  * Normal 7-10 point functionality
  * Moderate dysfunction of 4-6 points.
  * Severe dysfunction from 0 to 3 points.
Physical activity of the caregiver (BPAAT) | Baseline (at the start of the intervention) and at 12 months of treatment.
  Physical activity questionnaire adapted version . It measures physical activity, physical exercise.The Brief Physical Activity Assessment Tool (BPAAT) are valid and reliable assessment tools to identify "inactive" patients in primary. Brief Physical Activity Assessment Tool.
  It is a questionnaire administered by the healthcare professional. It consists of 2 questions that measure the frequency and duration of AF at vigorous and moderate intensity during a "typical" week. The scoring system identifies 'sufficiently active' patients (perform 3 sessions/week of 20 min at vigorous intensity or 5 sessions/week of 30 min at moderate intensity or 5 sessions of any combination of moderate or vigorous FA) or "insufficiently active" (do not meet healthy AF recommendations) care.
blood pressure of the child (systolic blood pressure and diastolic blood pressure) | Baseline (at the start of the intervention) and at 12 months of treatment
  systolic blood pressure and diastolic blood pressure (mm Hg)
waist circumference of the child | Baseline (at the start of the intervention) and at 12 months of treatment
  waist circumference (cm)
Sex | Baseline (at the start of the intervention)
  Sex (Male/ Female)
Age | Baseline (at the start of the intervention)
  Age (date of birth)

OTHER OUTCOMES:
Other Variables of the boy or girl | Baseline (at the start of the intervention)
  Antecedents of 1st degree obesity (yes / no).
Level of studies and other sociocultural and economic variables and of the main caregiver | Baseline (at the start of the intervention)
  Level of studies and other sociocultural and economic variables
Number of sessions attended by the caregiver (in case of intervention group). | 12 months
  Number of sessions attended by the caregiver (in case of intervention group).
Variables of the professional / Health Center: Years of experience in Primary Care | Baseline (at the start of the intervention)
  Years of experience in Primary Care.
Mother's weight | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment
  Weight in kilograms
Father's weight | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment
  Weight in kilograms
BMI of the Mother | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment
  weight and height will be combined to report BMI in kg/m^2)
BMI of the Father | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment
  weight and height will be combined to report BMI in kg/m^2)
Mother's Height | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment
  height in meters
Father's Height | Baseline (at the start of the intervention) and at 4, 6 and 12 months of treatment
  height in meters
Sex (Male /female) of the main caregiver | Baseline (at the start of the intervention)
  Sex (Male /female),
Change stage of the main caregiver | Baseline (at the start of the intervention) and at 12 months of treatment
  precontemplation (no motivation to be active) contemplation (motivation to change in the next 6 months) preparation (It has planned changes in the next month) action (active adherence to behavior lasting less than 6 months) maintenance (adherence to an active lifestyle greater than 6 months)
  (It has planned changes in the next month)
  action maintenance
Variables of the professional / Health Center: Sex (Male/ Female) | Baseline (at the start of the intervention)
  Sex (Male/ Female)

CONTACTS AND LOCATIONS:
Locations (1):
- Gerencia Asistencial de Atención Primaria de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollands GJ, Carter P, Anwer S, King SE, Jebb SA, Ogilvie D, Shemilt I, Higgins JPT, Marteau TM. Altering the availability or proximity of food, alcohol, and tobacco products to change their selection and consumption. Cochrane Database Syst Rev. 2019 Sep 4;9(9):CD012573. doi: 10.1002/14651858.CD012573.pub3. PMID 31482606
- [Background] Brown T, Moore TH, Hooper L, Gao Y, Zayegh A, Ijaz S, Elwenspoek M, Foxen SC, Magee L, O'Malley C, Waters E, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2019 Jul 23;7(7):CD001871. doi: 10.1002/14651858.CD001871.pub4. PMID 31332776
- [Background] Muthuri SK, Onywera VO, Tremblay MS, Broyles ST, Chaput JP, Fogelholm M, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Sarmiento OL, Standage M, Tudor-Locke C, Zhao P, Church TS, Katzmarzyk PT; ISCOLE Research Group. Relationships between Parental Education and Overweight with Childhood Overweight and Physical Activity in 9-11 Year Old Children: Results from a 12-Country Study. PLoS One. 2016 Aug 24;11(8):e0147746. doi: 10.1371/journal.pone.0147746. eCollection 2016. PMID 27557132
- [Background] Bammann K, Peplies J, Pigeot I, Ahrens W. [IDEFICS: a multicenter European project on diet- and lifestyle-related disorders in children]. Med Klin (Munich). 2007 Mar 15;102(3):230-5. doi: 10.1007/s00063-007-1027-2. German. PMID 17345019
- [Background] McKey S, Heinen M, Mehegan J, Somerville R, Khalil H, Segurado R, Murrin C, Kelleher CC; Lifeways Cross-Generation Cohort Study Steering Group. Predictors of adults' body mass index and the association with index child's infant birth weight, in the Lifeways Cross-Generation Cohort Study of a thousand families in the Republic of Ireland. J Dev Orig Health Dis. 2017 Dec;8(6):649-657. doi: 10.1017/S2040174417000435. Epub 2017 Jun 22. PMID 28637529
- [Background] Setayeshgar S, Ekwaru JP, Maximova K, Majumdar SR, Storey KE, McGavock J, Veugelers PJ. Dietary intake and prospective changes in cardiometabolic risk factors in children and youth. Appl Physiol Nutr Metab. 2017 Jan;42(1):39-45. doi: 10.1139/apnm-2016-0215. Epub 2016 Dec 13. PMID 27959641
- [Background] Ogden CL, Flegal KM, Carroll MD, Johnson CL. Prevalence and trends in overweight among US children and adolescents, 1999-2000. JAMA. 2002 Oct 9;288(14):1728-32. doi: 10.1001/jama.288.14.1728. PMID 12365956
- [Background] Sharifi M, Franz C, Horan CM, Giles CM, Long MW, Ward ZJ, Resch SC, Marshall R, Gortmaker SL, Taveras EM. Cost-Effectiveness of a Clinical Childhood Obesity Intervention. Pediatrics. 2017 Nov;140(5):e20162998. doi: 10.1542/peds.2016-2998. PMID 29089403
- [Background] Singh AS, Mulder C, Twisk JW, van Mechelen W, Chinapaw MJ. Tracking of childhood overweight into adulthood: a systematic review of the literature. Obes Rev. 2008 Sep;9(5):474-88. doi: 10.1111/j.1467-789X.2008.00475.x. Epub 2008 Mar 5. PMID 18331423
- [Background] Wilfley DE, Saelens BE, Stein RI, Best JR, Kolko RP, Schechtman KB, Wallendorf M, Welch RR, Perri MG, Epstein LH. Dose, Content, and Mediators of Family-Based Treatment for Childhood Obesity: A Multisite Randomized Clinical Trial. JAMA Pediatr. 2017 Dec 1;171(12):1151-1159. doi: 10.1001/jamapediatrics.2017.2960. PMID 29084318
- [Background] Freedman DS, Mei Z, Srinivasan SR, Berenson GS, Dietz WH. Cardiovascular risk factors and excess adiposity among overweight children and adolescents: the Bogalusa Heart Study. J Pediatr. 2007 Jan;150(1):12-17.e2. doi: 10.1016/j.jpeds.2006.08.042. PMID 17188605
- [Background] Metcalf PA, Scragg RK, Stewart AW, Scott AJ. Design effects associated with dietary nutrient intakes from a clustered design of 1 to 14-year-old children. Eur J Clin Nutr. 2007 Sep;61(9):1064-71. doi: 10.1038/sj.ejcn.1602618. Epub 2007 Jan 31. PMID 17268420
- [Background] Robson SM, Bolling C, McCullough MB, Stough CO, Stark LJ. A Preschool Obesity Treatment Clinical Trial: Reasons Primary Care Providers Declined Referrals. J Pediatr. 2016 Oct;177:262-266.e1. doi: 10.1016/j.jpeds.2016.06.027. Epub 2016 Jul 22. PMID 27453375
- [Background] Baker S, Barlow S, Cochran W, Fuchs G, Klish W, Krebs N, Strauss R, Tershakovec A, Udall J. Overweight children and adolescents: a clinical report of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. J Pediatr Gastroenterol Nutr. 2005 May;40(5):533-43. doi: 10.1097/01.mpg.0000161147.16590.12. PMID 15861011
- [Background] Golan M, Kaufman V, Shahar DR. Childhood obesity treatment: targeting parents exclusively v. parents and children. Br J Nutr. 2006 May;95(5):1008-15. doi: 10.1079/bjn20061757. PMID 16611394
- [Background] Epstein LH, Roemmich JN, Stein RI, Paluch RA, Kilanowski CK. The challenge of identifying behavioral alternatives to food: clinic and field studies. Ann Behav Med. 2005 Dec;30(3):201-9. doi: 10.1207/s15324796abm3003_4. PMID 16336071
- [Background] Rodearmel SJ, Wyatt HR, Stroebele N, Smith SM, Ogden LG, Hill JO. Small changes in dietary sugar and physical activity as an approach to preventing excessive weight gain: the America on the Move family study. Pediatrics. 2007 Oct;120(4):e869-79. doi: 10.1542/peds.2006-2927. PMID 17908743
- [Background] McGarvey E, Keller A, Forrester M, Williams E, Seward D, Suttle DE. Feasibility and benefits of a parent-focused preschool child obesity intervention. Am J Public Health. 2004 Sep;94(9):1490-5. doi: 10.2105/ajph.94.9.1490. PMID 15333300